CLINICAL TRIAL: NCT06175884
Title: Effectiveness of Physiotherapist's Communication Skills on Clinical Outcomes in Patients With Chronic Musculoskeletal Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of Physiotherapist's Communication Skills on Clinical Outcomes in Chronic Musculoskeletal Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantina Savvoulidou, Principal Investigator, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2023-11-27; First posted 2023-12-19 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: communication skills; chronic musculoskeletal pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Good communication skills (Experimental): Participants will watch a video about the pain neuroscience education in which physiotherapist will develop qualities of good communication while he will be giving information and explanation about chronic musculoskeletal pain.
  Interventions: Other: Video about pain neuroscience education with enhancing communication skills
- Poor communication skills (Experimental): Participants will watch a video about the pain neuroscience education in which physiotherapist will not develop qualities of good communication while he will be giving information and explanation about chronic musculoskeletal pain.
  Interventions: Other: Video about pain neuroscience education without enhancing communication skills
- Control (No Intervention): Participants will not watch any video

INTERVENTIONS:
Other: Video about pain neuroscience education with enhancing communication skills — Participants will watch a brief video on pain neuroscience in which physiotherapist will show evidence-based communication skills to effectively convey information to patients.
  Arms: Good communication skills
Other: Video about pain neuroscience education without enhancing communication skills — Participants will watch a brief video on pain neuroscience in which physiotherapist will not show evidence-based communication skills to effectively convey information to patients.
  Arms: Poor communication skills

SUMMARY:
The purpose of this study is to investigate the impact of the physiotherapist's communication on the clinical presentation of patients with chronic musculoskeletal pain.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the impact of the physiotherapist's communication on the clinical presentation of patients with chronic musculoskeletal pain. Sixty-nine (69) patients with chronic musculoskeletal pain in the cervical or lumbar spine, knee, or shoulder will participate. They will be randomly divided into three groups, each consisting of thirty-three (33) patients. One group (Experimental- Good communication skills) will watch the video in which physiotherapist will develop qualities of good communication while he explains about chronic musculoskeletal pain, the other group (Experimental- Poor communication skills ) will view the video in which the physiotherapist imparts information and explains chronic pain without enhancing his communication skills and lastly, the control group (control) that will not view any video.

ELIGIBILITY:
Inclusion Criteria:

* Participants should speak and understand the Greek language, as the questionnaires and the video will be in Greek
* Participants should experience pain in one of the following four different areas: cervical or lumbar spine, knee, or shoulder
* Pain of musculoskeletal origin
* Pain lasting more than 3 months, evident on most days of the week to be classified as chronic pain, with a pain intensity of at least 3/10 Numeric Pain Rating Scale.

Exclusion Criteria:

* Medication for neurological/psychiatric disorders
* Pain medication on the day agreed upon with the researcher, in order to minimize the potential influence of medication
* Undergoing surgery in the last six months
* Pregnancy or childbirth before 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
NPRS: Numeric Pain Rating Scale | Changes from baseline to10 minutes after watching the video
  The Numeric Pain Rating Scale will be utilized to evaluate the severity of pain. Participants will provide a score ranging from 0 (indicating no pain) to 10 (representing the most intense pain they have ever felt).
PPT: Pressure Pain Threshold | Changes from baseline to10 minutes after watching the video
  The Pain Pressure Threshold (PPT) is a method utilized to quantify the sensitivity of deep muscular tissues. In this measurement, an algometer is commonly employed to apply pressure to a specific area, and the point at which a gradually increasing pressure becomes painful is noted. In the context of PPT, lower values are indicative of heightened sensitivity, suggesting that the individual experiences pain at a lower pressure threshold. Therefore, lower PPT values are interpreted as an indication of increased sensitivity in the deep muscular tissues.

SECONDARY OUTCOMES:
Pain Distribution | Changes from baseline to10 minutes after watching the video
  The Pain Distribution App (PDA) will be employed to document the location of pain. This self-reported tool is designed to evaluate the distribution and extent of pain across different areas of the body. The reliability of the PDA has been previously demonstrated.
CSI: Central Sensitisation Inventory | Baseline
  The Central Sensitisation Inventory (CSI) serves as a self-report tool aimed at identifying individuals with symptoms potentially linked to Central Sensitisation. The inventory consists of two parts. Part A involves 25 questions related to common Central Sensitisation Syndrome (CSS) symptoms. Patients rate each question on a scale from 0 (never) to 4 (always). A total score exceeding 40 suggests the presence of central sensitisation. In Part B, patients indicate if they have received a diagnosis for specific CSS disorders or related conditions, such as anxiety and depression. Notably, only the scores from Part A are considered in the assessment.
BIPQ: Brief Illness Perception Questionnaire | Changes from baseline to 10 minutes after watching the video
  The Brief Illness Perception Questionnaire (B-IPQ) functions as an assessment tool for examining cognitive and emotional perceptions of illness. Comprising eight items, this questionnaire evaluates cognitive illness representation, emotional illness representation, and illness comprehensibility representation. Scoring involves rating each item on a scale from 0 to 10, where higher scores signify a more threatening perception of the illness. The total B-IPQ score is obtained by summing the scores of all eight items, resulting in a potential range of 0 to 80. Elevated scores on this scale indicate a more negative or distressing perception of the illness.
PCS: Pain Catastrophizing Scale | Changes from baseline to 10 minutes after watching the video
  The 13-item scale is structured around three dimensions: rumination over pain, magnification of pain, and helplessness in the face of pain symptoms. Both the total score and subscale scores for the Pain Catastrophizing Scale (PCS) are calculated by adding up the ratings for each item. In this study, the focus is on the total score, which ranges from 0 to 52, with higher scores indicating a higher level of pain catastrophizing.
STAI-40: State - Trait Anxiety Inventory | Changes from baseline to 10 minutes after watching the video
  The State-Trait Anxiety Inventory (STAI) is a psychological assessment tool comprising 40 self-report items, rated on a 4-point Likert scale. This inventory is designed to gauge two distinct forms of anxiety: state anxiety and trait anxiety. Elevated scores on the STAI are positively associated with increased levels of anxiety.
TSK: Tampa Scale for Kinesiophobia | Changes from baseline to 10 minutes after watching the video
  This questionnaire serves as a tool for assessing the fear of movement or the fear of (re)injury in individuals experiencing pain. The resulting score can range from a minimum of 11 to a maximum of 44 points, with a higher score indicating a greater degree of kinesiophobia. A score of ≥18 is considered indicative of a fear of movement, and the severity of this fear escalates with higher scores.
VES: Video Engagement Scale | Changes from baseline to 10 minutes after watching the video
  Video Engagement was evaluated using the Video Engagement Scale (VES-sf). This questionnaire, designed to measure participants' engagement while watching a video, consists of eight items rated on a scale from 0 ('totally disagree') to 7 ('totally agree'). Scores on the VES-sf range from 0 to 56, with higher scores indicating greater engagement during video viewing. To determine participant inclusion or exclusion, the specific item 'I was fully concentrated on the video while watching' was utilized. Participants with a score lower than 3 on this item were excluded from the study.
Working Alliance Inventory - Short Revised (WAI-SR) | Changes from baseline to 10 minutes after watching the video
  The measurement of bonding in the context of patient-physiotherapist interactions is conducted using the Bonding scale of the Working Alliance Inventory - Short Revised (WAI-SR). Bonding, a crucial component of the working alliance, is defined as the collaborative, warm, and supportive connection between a patient and a therapist. The WAI-SR bond scale assesses the quality of this bond and comprises four items, each rated on a scale from 1 ('never') to 5 ('always'). Scores on the bond scale range from 4 to 20, with higher scores indicative of a higher perceived quality in the bond between the patient and the therapist.
Global Rating of Change Scales | Changes from baseline to 10 minutes after watching the video
  The Global Rating of Change (GRoC) is a scale designed to evaluate the extent to which a patient's condition has improved, worsened, or remained stable, usually after receiving treatment. The GRoC typically involves a single question that prompts the patient to rate the change in their specific condition over a defined time frame. The GRoC is an 11-point scale, ranging from -5 (indicating a significant deterioration or being "very much worse") to 0 (representing no change or "unchanged") and up to +5 (indicating complete recovery or being "completely recovered").

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Kapreli, Study Chair — University of Thessaly
Locations (1):
- University of Thessaly, Lamia, Greece

IPD SHARING:
Plan to Share IPD: No